CLINICAL TRIAL: NCT00003508
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Patients With Mesothelioma
Brief Title: Antineoplaston Therapy in Treating Patients With Advanced Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to slow enrollment
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066551; BC-MA-2 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-01

CONDITIONS: Malignant Mesothelioma
Keywords: advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm: Experimental: Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with advanced mesothelioma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.hourly interEach infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for advanced Mesothelioma provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of advanced Mesothelioma.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with advanced Mesothelioma.

DETAILED DESCRIPTION:
Advanced Mesothelioma patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with advanced Mesothelioma, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with advanced Mesothelioma.
* To determine objective response, tumor size is measured utilizing physical examination and radiologic studies, performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV mesothelioma that is unlikely to respond to existing therapy and for which no curative therapy exists

  * Evidence of disease by CT scan or MRI

PATIENT CHARACTERISTICS:

Age:

* 1 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal
* Hepatic function adequate

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal insufficiency
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension
* No history of congestive heart failure
* No cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No serious lung disease (e.g., chronic obstructive pulmonary disease)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* Not at high medical or psychiatric risk
* No nonmalignant systemic disease
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulatory agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy (or less if multiple tumors) and recovered

Surgery:

* Recovered from prior surgery

Other:

* Prior cytodifferentiating agents allowed
* No prior antineoplastons
* No other concurrent antineoplastic agents

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1996-03-08 (Actual); Primary Completion 2005-04-26 (Actual); Study Completion 2005-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Study Chair — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Preliminary findings on the use of targeted therapy in combination with sodium phenylbutyrate in advanced malignant mesothelioma: A strategy for improved survival. Journal of Cancer Therapy. 2014; 5:1127-1144.
- [Background] Burzynski SR, Lewy RI, Axler M, Janicki TJ.Treatment of malignant mesothelioma (MM) with sodium phenylbutyrate.Presented at the 15th International Congress on Anti-Cancer Treatment; February 9-12, 2004, Paris, France.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm: Experimental: Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Patients with advanced mesothelioma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.hourly interEach infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Period: Overall Study
Arm/Group | Arm: Experimental: Antineoplaston Therapy
Started | 8
Completed | 3
Not Completed | 5
Not completed — Not evaluable | 5

BASELINE CHARACTERISTICS:
Population: Eight patients were enrolled in the study, only 3 patient was evaluable.
Units Other Than Participants: Evaluable Patients
Arm/Group | Arm: Experimental: Antineoplaston Therapy
Number analyzed (Participants) | 8
Number analyzed (Evaluable Patients) | 3
Age, Continuous [Median (Standard Deviation); unit: years] | 60.0 (8.9527)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response, Stable Disease, Progressive Disease or Not Evaluable
Description: Objective response rate per The International Working Group response criteria (1999): Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable lesions, sustained for at least four weeks. Stable Disease (SD), < 50% change in the sum of the products of of the greatest perpendicular diameters of all measurable lesions, sustained for at least twelve weeks.
Time Frame: 109 months
Population: All patients enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Arm: Experimental: Antineoplaston Therapy
Number analyzed (Participants) | 8
participants
  Objective Response | 0
  Stable Disease | 2
  Progressive Disease | 1
  Not evaluable | 5

ADVERSE EVENTS:
Time Frame: 9 years, 1 month
Description: Eight patients were recruited between March 1966 and April 2005. All study subjects were seen at the Burzynski Clinic in Houston TX.
Arm/Group | Arm: Experimental: Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm: Experimental: Antineoplaston Therapy (N=8)
Hemorrhage, pulmonary: Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1
Infection NOS (Infections and infestations) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm: Experimental: Antineoplaston Therapy (N=8)
Allergic reaction/hypersensitivity (including drug fever) (General disorders) | 2
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (General disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Hypertension (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Central Venous Catheter Infection (Infections and infestations) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5
Fever (General disorders) | 1
Rigors/chills (General disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 3
Cushingoid appearance (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1
Hemorrhage, pulmonary: Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary: Nose (Respiratory, thoracic and mediastinal disorders) | 1
Infection (Infections and infestations) | 1
Infection (documented clinically): Bronchus (Infections and infestations) | 1
Infection (documented clinically): Skin (cellulitis) (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 2
Alkaline phosphatase (Investigations) | 2
Hyperglycemia (Investigations) | 1
Hyperkalemia (Investigations) | 1
Hypernatremia (Investigations) | 4
Hypocalcemia (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No